CLINICAL TRIAL: NCT04282265
Title: The Effects of Red Spinach Extract on Health on Physical Performance Following Chronic Resistance Training in Trained Males
Brief Title: The Effects of Red Spinach Extract on Physical Performance Following Chronic Resistance Training in Trained Males
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Lipscomb University (Other)
Responsible Party: Principal Investigator, Jeremy Townsend, Assistant Professor, Lipscomb University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: 050719
Record Dates: First submitted 2020-01-16; First posted 2020-02-24 (Actual); Last update posted 2020-02-24 (Actual); Status verified 2020-02

CONDITIONS: Sports

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Placebo (Placebo Comparator)
  Interventions: Dietary Supplement: Placebo
- Red Spinach Extract (Experimental)
  Interventions: Dietary Supplement: Red Spinach Extract (RSE)

INTERVENTIONS:
Dietary Supplement: Placebo — Oral placebo capsules will be taken consisting of maltodrextrin daily for 11 weeks
  Arms: Placebo
Dietary Supplement: Red Spinach Extract (RSE) — Oral capsules containing 2g of Red Spinach Extract will be consumed daily for 11 weeks
  Arms: Red Spinach Extract

SUMMARY:
Red Spinach is a natural food which is a rich source of nitrates, which are beneficial in hemodynamics, cardiovascular function, and have natural hypotensive and antianginal effects . In recent research, Red spinach extract has been shown to be beneficial in acute exercise performance. However, currently it is unclear how these acute increases in performance may translate to long term training adaptations.

This research study is designed to measure the effects of red spinach extract (RSE) on markers of physical performance, body composition, and health following chronic resistance training and anaerobic exercise.

DETAILED DESCRIPTION:
The investigators aim to measure muscle strength, athletic performance, body composition, and muscle size in two groups of adults before and after 11 weeks of intervention in a randomized, double blinded study. One group (n=15 ) will receive an intervention of resistance exercise and a Red Spinach Extract supplement, and the other group (n=15) will receive resistance exercise and a placebo (maltodextrin).

ELIGIBILITY:
Inclusion Criteria:

* 18-35 years old
* At least 1 year of resistance training experience
* Are free of musculoskeletal injuries
* Are not taking medications that may interfere with study measurements

Exclusion Criteria:

* Participant that cannot take either the RSE or placebo supplement will be excluded, as this will be a double-blind study.
* Furthermore, participants that cannot participate in pre- and post-research testing, and/or those that cannot commit to regular training sessions will be excluded.
* Inability to perform physical exercise (determined by health and activity questionnaire)
* Taking any other nutritional supplement or performance enhancing drug.
* Any chronic illness that causes continuous medical care.

Ages: 18 Years to 34 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2019-08-23 (Actual); Primary Completion 2019-11-29 (Actual); Study Completion 2019-11-29 (Actual)

PRIMARY OUTCOMES:
Muscular Strength | 11 weeks
  Muscular strength will be assessed via bench press 1-repetition maximum
Muscular Hypertrophy | 11 weeks
  Muscle thickness of the Rectus femoris and vastus lateralis will be assessed via ultrasonography. Thickeness will be reported in cm.
Body Composition | 11 weeks
  Lean Body Mass, Fat Mass, and Bone Mineral Content will be assessed via Dual X-ray absorptiometry (DXA)
Wingate Anaerobic (WnT) Cycle test performance | 11 weeks
  A 30-second WnT test will be used to assess Average power, peak power, and fatiuge index

CONTACTS AND LOCATIONS:
Locations (1):
- Jeremy Townsend, Nashville, Tennessee, United States